CLINICAL TRIAL: NCT05858502
Title: Understanding the Determinants of Mucosal Immunity and Optimizing the Diagnosis of Infection With SARS-CoV-2 Variants
Acronym: COVARIANT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Biogroup Laboratoire de biologie médicale (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-079; 2022-A02703-40 (Other: ID-RCB)
Record Dates: First submitted 2023-05-12; First posted 2023-05-15 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Blood sample collection — Blood sample collection between inclusion and 3 months max 55 ml at each visit
Other: Saliva sample collection — Saliva sample collection between inclusion and 3 months
Other: Nasopharyngeal and nasal sample collection — Nasopharyngeal and nasal sample collection between inclusion and 3 months
Other: Exhaled Breath Condensate (EBC) — Exhaled Breath Condensate (EBC) between inclusion and 3 months

SUMMARY:
One of the current health challenges in the face of the COVID-19 pandemic that started in Wuhan in 2019, and still responsible for successive waves, is to better understand and diagnose the infection.

The new variants - delta, then omicron, which appeared in November 2021 and then their sub-variants BA.2, then BA.4 and 5, and more recently BQ.1 and the sub-variant XBB.1.5 are increasingly transmissible and responsible for some degree of immune escape. Hence the importance of a better understanding of infection- or vaccine-induced immunity in order to optimize existing prophylactic or therapeutic strategies, or even to develop new, more effective ones.

Mucosal immunity could play a particularly important role in interrupting the infection cycle at the entry point of the virus.

The key role of innate immunity has been demonstrated in particular, via interferons and the composition of the microbiota.

Humoral immunity is the best documented. However, it tends to be eroded within a few months. On the other hand, cellular immunity is more stable over time and would largely explain the decrease in severe forms of the disease in vaccinated individuals.

The collection of biological resources that will be built up during this study will also allow us to optimize or develop new diagnostic methods, necessary as a complement to vaccination, to effectively slow down the spread of the pandemic and reduce the severity of its impact on the population.

The improvement of diagnostic methods will in turn improve the understanding of the infection by providing increasingly reliable information on the characteristics of an infection, its quantification, its dynamics, and its resolution, especially since these parameters will be compared, at any time during the study, with reference methods and the immunological status of the subject.

The main significant improvements expected in the field of SARS-CoV-2 diagnosis are notably the improvement of performance (reduction of false negatives in RT-PCR on nasopharyngeal samples), acceptability, simplicity of implementation in the field, and the capacity to test transmission.

The objective of this study is to identify and characterize SARS-CoV-2 infection and host response, particularly mucosal immunity.

DETAILED DESCRIPTION:
This is a prospective, longitudinal, descriptive study that will include adult participants infected and uninfected with Sars-CoV-2 at the time of recruitment.

Participants will be divided into 3 groups of 30 evaluable subjects:

* uninfected,
* asymptomatically infected,
* symptomatically infected.

The participants will be identified within the Ile-de-France medical analysis laboratories partners of the project.

Study with sample collection:

- For participants infected with SARS-CoV-2: Inclusion visit V0, ≤ 3 days after PCR test Follow-up visit V1, 7 d ± 1 d after V0 Follow-up visit V2, 31 d ± 2 d after V0 V3 follow-up visit, 91 d ± 5 d after V0

- For participants not infected with SARS-CoV-2 : Inclusion visit V0, ≤ 3 days after PCR test V1' visit, no more than 96 d after V0.

ELIGIBILITY:
Inclusion Criteria:

* Common criteria for all subjects:

  * Aged between 18 and 65 years included
  * Whose weight is greater than or equal to 50 kg and whose state of health is compatible with the collection of 55 ml of blood at one time and 111 ml in 28 days
  * Residing in the Ile-de-France region and able to travel to the 15th arrondissement of Paris for visits to ICAReB-Clin
  * Having given their consent to participate in the study
  * Benefiting from a Social Security scheme except for the Aide Médicale d'Etat
* Criteria for the SARS-CoV-2 infected participant group:

  * Subject tested positive for SARS-CoV-2 by RT-PCR in one of the participating laboratories for less than 72 hours
  * Asymptomatic or with symptoms not requiring hospitalization regardless of previous vaccination or infection status for SARS-CoV-2.
* Criteria for the SARS-CoV-2 uninfected group:

  * Having tested negative for SARS-CoV-2 by RT-PCR
  * Subject with no more than 3 co-morbidities listed by the HAS.

Exclusion Criteria:

* Criteria common to all subjects :

  * Subject under a protective measure (e.g., guardianship)
  * Participant in another biomedical research
  * For women: pregnant or breastfeeding women (declarative)
  * Subject with another acute infectious disease
  * SARS-CoV-2 RT-PCR result older than 3 days
  * Existence of at least 3 co-morbidities known to be factors of severity (and therefore representing risks of hospitalisation during follow-up)
  * Existence of a previous known SARS-CoV-2 positivity less than 1 month old (whatever the method used: RT-PCR or antigenic test)
* SARS-CoV-2 infected participant group criteria:

  - For symptomatic subjects: onset of symptoms more than 4 days ago
* SARS-CoV-2 uninfected participant group criteria:

  * Known history of infection and/or COVID-19 vaccination, within the previous 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
To characterize SARS-CoV-2 infection and host response, particularly mucosal immunity. | 12 months
  Measurement of mucosal anti-SARS-CoV-2 antibody levels and cytokines, composition of the local microbiota of the upper respiratory tract.

SECONDARY OUTCOMES:
To characterize biomarkers of infection (stage, severity, prognosis) with new innovative direct or indirect diagnostic methods for SARS-CoV-2 and identify potential theranostic biomarkers. | 12 months
  Measurement of the capacity of the biomarkers to characterize the different stages, severity and prognosis of the infection, or theranostic potential.
To characterize the dynamics of infection and immunological response from the date of suspected infection and up to 3 months post-infection, or later, during the first year | 12 months
  Kinetics of virological evolution and immune response in different compartments (blood, upper and lower respiratory)
To develop tools to assess the contamination capacity of subjects. | 12 months
  Measurement of viral load in exhaled air condensates
To characterization of mucosal and humoral immunity. | 12 months
  Measurement and comparison of mucosal and humoral immunity parameters
To optimize sampling techniques and calibrate the detection of viral components by artificial contamination on samples taken during the 1st visit of uninfected subjects. | 12 months
  Measurement of viral detection calibration results on the 1st visit samples of uninfected subjects

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Laude, MD, Principal Investigator — Institut Pasteur
Locations (1):
- Institut Pasteur - ICAReB-clin, Paris, France

IPD SHARING:
Plan to Share IPD: No